CLINICAL TRIAL: NCT03491137
Title: Wireless Assessment of Respiratory and Circulatory Distress in Surgical Patients
Brief Title: Wireless Assessment of Respiratory and Circulatory Distress
Acronym: WARD
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Technical University of Denmark (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Camilla Haahr-Raunkjær, MD, principal investigator, Bispebjerg Hospital
Other Study IDs: H-17033535
Record Dates: First submitted 2018-01-30; First posted 2018-04-09 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Complications
Keywords: Wireless monitoring, postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A high percentage of patients undergoing major abdominal surgery will develop a postoperative complication. Our hypothesis is that by observing postoperative patients with continuous wireless monitoring, it is possible to detect the correlation between deviating vital parameters and subsequent postoperative complications. A prospective observational study will take place on general surgical wards with the enrolment of 500 patients in two different hospitals. Physiological parameters will be recorded for 96 hours postoperative. Data is collected preoperative, peroperative and postoperative in up to 6 months for data analyzing.

DETAILED DESCRIPTION:
An estimated > 230 million cases of major surgery are performed worldwide annually. Surgical interventions come with an inherent risk of complications. 15 - 30 % of all patients undergoing major abdominal surgery will develop a severe complication post-operative. These numbers correspond to the reported high postoperative in-hospital mortality, 8-9% after major upper abdominal surgery, increased in case of co-morbidities. Part of the high morbidity and mortality may be a result of delayed detection of severe complications due to the lower monitoring frequency in the general wards compared to the Post Anaesthesia Care Unit (PACU) and Intensive Care Unit (ICU). Improved observation may result in earlier detection and subsequently the possibility to implement interventions to divert a negative trajectory and ultimately reduce morbidity and mortality.

This study wish to investigate the correlation between deviating physiological parameters and postoperative complications.

In a prospective observational study, 500 patients enrolled for major abdominal cancer surgery at Rigshospitalet or Bispebjerg Hospital will be included after a signed declaration of consent.

Demographic data will be recorded together with preoperative spirometry, timed-up-and-go, Mini Mental State Examination and an electrocardiogram.

Post-operative when leaving the PACU, a wireless continuous monitoring system will be attached to the patients. The monitoring system will be recording the vital parameters 24/7.

In parallel to the wireless monitoring, the patients will receive normal treatment and monitoring (Early Warning Score) from staff on the wards. Patients are monitored for 96 hours or until they are dismissed from hospital.

Furthermore blood samples will be collected once every day for 96 hours and the patients are appointed daily by an investigator.

Exposure variables is deviation of vital parameters from normal range, socalled microevents.

Descriptive statistic will be used in analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 60 years old
* Elective operation performed at Bispebjerg Hospital or Rigshospitalet.
* Elective major abdominal cancer surgery.
* Operation estimated to last more than 2 hours.

Exclusion Criteria:

* Mortality.
* Non-cooperative patients.
* Patients with mini mental state examination score < 24.
* Patients allergic to plaster or silicone.
* Patients with ICD or pacemaker

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled for elective abdominal cancer surgery at Bispebjerg Hospital or Rigshospitalet will be invited to be a part of this study if they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Any serious adverse event | within 30 days after inclusion
  e.g cardiac arrest, ICU admission, acute myocardial infarction, sepsis, stroke, acute kidney injury, pneumonia or other serious adverse events (defined in Protocol Appendix A)

SECONDARY OUTCOMES:
Mortality | 6 months postoperative
Readmission | 6 months postoperative
  Acute readmission to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Haahr-Raunkjær, MD, Principal Investigator — Surgical department, Bispebjerg Hospital; Eske K Aasvang, Dr.med., Study Chair — Abdominal surgical department, Rigshospitalet
Locations (2):
- Denmark (2):
  - Abdominal surgical department, Rigshospitalet, Copenhagen
  - Surgical department, Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No
No plan of sharing IPD to other researchers

REFERENCES:
- [Derived] Jokinen JDV, Carlsson CJ, Rasmussen SM, Nielsen OW, Winkel BG, Jorgensen LN, Achiam MP, Molgaard J, Sorensen HBD, Aasvang EK, Meyhoff CS; WARD Project Group. Wireless Single-Lead ECG Monitoring to Detect New-Onset Postoperative Atrial Fibrillation in Patients After Major Noncardiac Surgery: A Prospective Observational Study. Anesth Analg. 2022 Jul 1;135(1):100-109. doi: 10.1213/ANE.0000000000005960. Epub 2022 Feb 25. PMID 35213523
- [Derived] Haahr-Raunkjaer C, Molgaard J, Elvekjaer M, Rasmussen SM, Achiam MP, Jorgensen LN, Sogaard MIV, Gronbaek KK, Oxboll AB, Sorensen HBD, Meyhoff CS, Aasvang EK. Continuous monitoring of vital sign abnormalities; association to clinical complications in 500 postoperative patients. Acta Anaesthesiol Scand. 2022 May;66(5):552-562. doi: 10.1111/aas.14048. Epub 2022 Feb 28. PMID 35170026